CLINICAL TRIAL: NCT04221139
Title: Virtual Reality: Its Effect on Physical Activity Intensity and Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kelly Naugle, PhD, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1907886495
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Physical Activity
Keywords: Virtual reality; active gaming; Physical activity; exercise-induced hypoalgesia
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy young adults (Experimental): Healthy young adults will play four virtual reality games: Beat Saber, Holopoint, Hot Squat, and Relax Walk.
  Interventions: Behavioral: Virtual Reality games

INTERVENTIONS:
Behavioral: Virtual Reality games — Participants will play the following four virtual reality games for 15 minutes each: Beat Saber, Holopoint, Hot Squat, and Relax Walk.

SUMMARY:
The purpose of this research study is to evaluate physical activity intensity levels, enjoyment, and pain perception during virtual reality (VR) active games in healthy young adults.

DETAILED DESCRIPTION:
Enrolled participants will complete four sessions: the first session including the informed consent process and one experimental game, and sessions 2-4 being devoted to one experimental game per session.

Screening and enrollment (Session 1 only): All participants will be asked to read and sign an Informed Consent Form (ICF) and a copy of the ICF will be given to the participant to keep for their records. Following the ICF process, participants will be given the Physical Activity Readiness-Questionnaire Plus (2019 version), a demographic questionnaire, and the International Physical Activity Questionnaire (IPAQ) to fill out. Inclusion and exclusion criteria will be assessed and eligibility will be determined.

Familiarization of pain test and VR system (Session 1 only):

Participants will undergo a familiarization with the pressure pain threshold (PPT) test to measure pain sensitivity. The PPT test will be performed as practice on the participants' non-dominant forearm and thigh three times. Following PPT familiarization, participants will be shown the HTC Vive system, which includes a head-mounted display system and two handheld controllers. The HTC Vive system comes with a tutorial program which exposes the user to the basic functions of the VR system. Each participant will be fitted with the headset and follow the tutorial for movement/system familiarization.

Experimental Protocol (All sessions): In each session participants will play one of the following four virtual reality games: Beat Saber, Holopoint, Hot Squat, and Relax Walk. The order of the games played in Sessions 1 - 4 will be randomized and counterbalanced. Following the familiarization via the tutorial program (only Session 1), participants will be introduced to one of the games (which will be randomized). A verbal description of the game followed by a visual demonstration will be conducted by the researcher for the participant to observe. The participant will then play the game for approximately 10 minutes for familiarization. After 10 minutes, the participants will be asked to stop playing and sit in a resting position to allow for a proper return to resting heart rate.

Participants will wear accelerometers on the hip and arm to measure physical activity behavior during game play. Participants will also wear heart rate monitors during game play. The participants will then play the game for 15 minutes. Every 5 minutes the participant will be asked to rate their exertion using the Borg 6-20 Ratings of Perceived Exertion (RPE) scale. After 15 minutes of game play, the pressure pain thresholds will be administered on the leg and forearm. The participant will then be allowed/assisted in removing the VR headset and will be asked to rate their level of enjoyment using an 11-point Visual Analog Scale. The next session will be scheduled with the participant. Session 1 is expected to last 1.5 hours and sessions 2 through 4 will last approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 30 years old.

Exclusion Criteria:

* Prior or current events with motion sickness or claustrophobia
* Any acute or chronic pain condition
* If "yes" is answered on any of the general health questions on the Physical Activity Readiness Questionnaire (PAR-Q+ 2019 version) and the subsequent answer of "yes" on any follow-up question on the about any present medical condition will exclude a participant. The initial seven questions on the form include the following with more extensive follow-up questions in the event that any are answered with "yes."

  * If participant's doctor has ever said that he/she has a heart condition and that he/she should only do physical activity recommended by a doctor
  * Pain in chest when doing physical activity
  * In past month, chest pain when not doing physical activity
  * If participant has ever lost balance because of dizziness or has ever lost consciousness
  * Bone or joint problem that could be made worse by change in physical activity
  * Currently on prescribed drugs for blood pressure or heart condition.
  * If the participant knows of any other reason why he/she should not do physical activity.

Session exclusion criteria:

* Severe uncontrolled hypertension: resting Systolic blood pressure > 180mmHg, resting diastolic blood pressure> 99mmhg
* Participating in vigorous exercise at least 12 hours prior to study sessions, eating at least 1 hour prior to each session, and smoking, consuming alcohol for 24 hours, and caffeine, and analgesic medications on the day of the session prior to the session.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Ratings of perceived exertion | This measure will be assessed immediately after playing the virtual reality games
  Ratings of Perceived Exertion Borg Scale. The minimum value is 6, indicating no exertion. The maximum value is 20, indicating maximal exertion.
Whole body percentage of time spent in moderate to vigorous physical activity | This measure will be assessed during the 15 minutes of each virtual reality game play.
  Participants will wear an accelerometer on the hip during the virtual reality games. Activity count cut points can identify the amount of time spent in moderate to vigorous physical activity during game play.
Arm percentage of time spent in moderate to vigorous physical activity | This measure will be assessed during the 15 minutes of each virtual reality game play.
  Participants will wear an accelerometer on the dominant arm during the virtual reality games. Activity count cut points can identify the amount of time spent in moderate to vigorous physical activity during game play.
Whole body Percentage of time spent in sedentary time | This measure will be assessed during the 15 minutes of each virtual reality game play.
  Participants will wear an accelerometer on the hip during the virtual reality games. Activity count cut points can identify the amount of time spent in sedentary behavior during game play.
Arm percentage of time spent in sedentary time | This measure will be assessed during the 15 minutes of each virtual reality game play.
  Participants will wear an accelerometer on the dominant arm during the virtual reality games. Activity count cut points can identify the amount of time spent in sedentary behavior during game play.
Average percentage of heart rate reserve during game play | This measure will be assessed during the 15 minutes of each virtual reality game play.
  Participants will be fitted with a Polar heart rate monitor (Polar Electro) at the beginning of each experimental session and will be monitored during gameplay. Heart rate values will be used to calculate percentages of heart rate reserve (HRR) for interpreting intensity levels.

SECONDARY OUTCOMES:
Enjoyment | This measure will be assessed immediately after each virtual reality game is played.
  participants will be asked to complete an 11-point visual analogue scale indicating their level of enjoyment while playing the active game, with 0 indicating no enjoyment and 10 indicating the most enjoyment one could experience.
Enjoyment during game play | This measure will be assessed immediately after each virtual reality game is played.
  Participants will complete the modified Physical Activity Enjoyment Scale (PACES), which includes Likert-style questions asking about enjoyment during physical activity. The score ranges from 5 to 35, with a higher value indicating higher enjoyment.
Pressure pain sensitivity | This measure will be assessed before the virtual reality games and immediately after the virtual reality games are played.
  Using a hand-held, clinical grade pressure algometer (Wagner Instruments, Greenwich, CT), pressure will be applied to the dominant forearm and thigh. Pressure will increase at a rate of about 1kg/s until the subject first reports feeling pain.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Fitness and Sport, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Evans E, Naugle KE, Kaleth AS, Arnold B, Naugle KM. Physical Activity Intensity, Perceived Exertion, and Enjoyment During Head-Mounted Display Virtual Reality Games. Games Health J. 2021 Oct;10(5):314-320. doi: 10.1089/g4h.2021.0036. Epub 2021 Aug 27. PMID 34449262